CLINICAL TRIAL: NCT03633318
Title: Application of Electrical Impedance Myography (EIM) to Establish Muscle Impedance Parameters as a Potential Biomarker of Inclusion Body Myositis (IBM)
Brief Title: Establishing Muscle Impedance Parameters With Electrical Impedance Myography
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000023035
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: IBM; Inclusion Body Myositis
Keywords: electrical impedance myography; EIM
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- IBM Group: Participants in this arm will have Inclusion Body Myositis (IBM). All patients will have EIM measurements of selected muscles.
  Interventions: Device: electrical impedance myography (EIM)
- Control Group: Participants in this arm will be healthy controls. All participants will have EIM measurements of selected muscles.
  Interventions: Device: electrical impedance myography (EIM)

INTERVENTIONS:
Device: electrical impedance myography (EIM) — EIM is a measure of impedance. EIM is a measure of the obstruction of flow of current through the tissue. It is a completely painless assessment of muscle health.

SUMMARY:
The primary aim of this study is to assess the changes in the impedance parameters of muscles in inclusion body myositis (IBM) through electrical impedance myography (EIM), an emerging non-invasive electrodiagnostic technology. Muscle impedance parameters can potentially serve as an objective biomarker reflecting disease progression and severity.

DETAILED DESCRIPTION:
In this pilot study, the electrical impedance myography (EIM) parameters of individuals with inclusion body myositis (IBM) will be compared with age and sex matched normal data. Along with EIM parameters, clinical outcome measures will be obtained to understand how EIM data correlates with these parameters. A focused study to assess muscle health in IBM patients through EIM is essential to gather further insight into the potential application of this technology as a disease biomarker. Additionally, this investigation will provide critical data for the design of a subsequent biomarker validation study.

ELIGIBILITY:
Inclusion Criteria:

* Clinico-pathologically defined IBM in the absence of any other significant neurological problem or cognitive dysfunction.
* Healthy controls will be age and gender-matched to the enrolled IBM patients.

Exclusion Criteria for both IBM and control group:

* Patients with decompensated congestive heart failure
* Patients with chronic kidney disease on hemodialysis
* Patients with active cancer on chemotherapy or radiotherapy
* Patients with severe disease who are already wheel-chair bound

Min Age: 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with IBM compared with age and sex matched people of typical health with: no active neuromuscular disorders or known history of neuromuscular disorders; no sign or symptoms of muscle weakness; no family history of muscular dystrophies or ALS.
  .
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
IBM-Functional Rating Scale | 45 Minutes
  Physical functioning in daily life will be measured using the IBM-Functional rating scale (IBM-FRS). IBM-FRS will be obtained for both IBM participants and healthy controls.
Grip Strength | 45 Minutes
  Grip strength will be assessed using the Jamar hand dynamometer and will be obtained by the physician from both IBM participants and healthy controls. The best of three attempts will be used.
Time to Stand | 45 Minutes
  Time to stand will be measured using the "Get-up-and-go test". Time will be measured for a participant to stand up from a chair (using arms if necessary), walk 3 meters, turn around, return to the chair, and sit down. The better of two trials will be used. These results will be obtained by the physician from both IBM participants and healthy controls.
Walking Distance | 45 Minutes
  Distance walked by a participant in 6 minutes will be measured. Given the general disability of many IBM participants, rather than utilizing two trials, a 2-minute "practice" walk will be performed before the actual test, to familiarize the participant with the task to be performed. Both IBM participants and healthy controls will undergo this procedure.
Manual Muscle Testing (MMT) Global Score | 45 Minutes
  This is a hands-on assessment that will use the Medical Research Council muscle scales (MRC) to score the strength of the following muscle groups that may be involved in IBM: neck flexor, extensor, deltoid, biceps, triceps, wrist extensor, wrist flexors, finger long and short flexors, finger extensors, hip flexors, hip adductors, hip abductors, knee extensors, knee flexors, ankle dorsi and planti flexors. MRC scores will be obtained by the physician from both IBM participants and healthy controls. A global score can be calculated and will be used. 0 (none) = no contraction, 1 (trace) = visible contraction with no motion, 2 (poor) = full range of motion, gravity eliminated, 3 (fair) = full range of motion against gravity, 4 (good) = full range of motion against gravity, moderate resistance, 5 (normal) = full range of motion against gravity, maximum resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Bhaskar Roy, MBBS, Principal Investigator — Yale School of Medicine: Department of Neurology; Richard J Nowak, MD, MS, Principal Investigator — Yale School of Medicine: Department of Neurology
Locations (1):
- Yale Physicians Building, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No